CLINICAL TRIAL: NCT04878614
Title: Comparison of Levothyroxine Formulation in Hypothyroid Patients With Enteral Feeding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated study low accrual numbers
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Vijaya Surampudi MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#20-002097
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Hypothyroidism
Keywords: Levothyroxine; Enteral Nutrition; Gastrostomy Tube
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial.
Who Masked: Participant
Masking Description: Participants will be randomized 1:1 to either continue current management with the same dose or to dose equivalent liquid levothyroxine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Levothyroxine Management (Active Comparator): Participants will continue with the same regimen
  Interventions: Drug: Levothyroxine Tablet
- Liquid Levothyroxine Management (Experimental): Participants will be treated with dose equivalent regimen through enteral feeding tube
  Interventions: Drug: Levothyroxine Sodium

INTERVENTIONS:
Drug: Levothyroxine Tablet — Standard clinical management
  Arms: Standard Levothyroxine Management
Drug: Levothyroxine Sodium — Liquid levothyroxine through enteral feeding tube
  Other Names: Tirosint-SOL
  Arms: Liquid Levothyroxine Management

SUMMARY:
The purpose of this study is to test a liquid levothyroxine formula and examine if it will lead to improvement in management of thyroid function and if it improves hypothyroid symptoms that patients experience.

DETAILED DESCRIPTION:
Patients who require enteral nutrition through an enteral feeding tube and have hypothyroidism often struggle with the management of hypothyroidism. Hypothyroidism usually requires lifelong treatment except in some cases. It has been clinically observed the traditional management of hypothyroidism is to crush the tablet and administer the medical through the enteral nutrition tube and hold the feeds for one hour. However, management of the hormonal profile has been noted to have variable results with this method. Limited data is available about the effectiveness of levothyroxine liquid formulation in outpatients' dependent on enteral feeding tubes for administration.

Therefore, we propose a study to assess if daily treatment of, Tirosint-SOL (liquid levothyroxine, IBSA pharma Inc.), will improve thyroid function tests in individuals requiring enteral nutrition and are hypothyroid in a prospective, randomized study in a population requiring enteral nutrition. We hypothesize that Tirosint-SOL will lead to improvement in management in their thyroid function tests resulting in possible improvement in hypothyroid symptoms experienced by the patients.

This will be a randomized controlled trial. The study will be conducted in patients who have uncontrolled hypothyroidism on levothyroxine therapy. These patients will also be dependent on enteral nutrition and medication administration through the gastrostomy tube. The participants will be followed at UCLA Enteral Nutrition Clinic. Participants will be randomized 1:1 to either continue current management with the same dose or to dose equivalent liquid levothyroxine. At baseline (week 0) and week 6-8, TSH and thyroid function tests will be performed. In addition, medical history and physical, body weight, HR, blood pressure, nutritional intake by a registered dietitian will be done at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years old or older
* G-tube/G-J tube dependent for medication administration
* Hypothyroid patients on levothyroxine tablet
* TSH>5 on levothyroxine

Exclusion Criteria:

* J-tube
* Unstable cardiac condition
* Unstable gastrointestinal condition
* Unable to reliably administer medication
* Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* In the opinion of the study investigator, any subject who demonstrate a risk of non-compliance with study procedure, or one who cannot read, understand or complete study - related materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change of TSH | 6 weeks
  evaluate change in thyroid hormonal panel

SECONDARY OUTCOMES:
percentage of patients with therapeutic FT4 | 6 weeks
  evaluate change in thyroid hormonal panel
percentage of patients with therapeutic FT3 | 6 weeks
  evaluate change in thyroid hormonal panel

CONTACTS AND LOCATIONS:
Overall Officials: Vijiya Surampudi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States